CLINICAL TRIAL: NCT06845735
Title: Prospective Randomized Control Trial Comparing Absorbable Sutures to Non-Absorbable Sutures for Capsular Closures in Hip Arthroscopies
Brief Title: Absorbable vs Non-Absorbable Sutures for Hip Capsular Closure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Steven DeFroda, Asst Prof Orthopaedic surgery, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2099469
Record Dates: First submitted 2025-01-27; First posted 2025-02-25 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Labrum Injury of the Hip Joint; Hip Arthroscopy; Femoroacetabular Impingement Syndrome
MeSH Terms: conditions — Femoracetabular Impingement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Absorbable Suture (Active Comparator): Absorbable suture
  Interventions: Device: Absorbable Suture
- Non-Absorbable Suture (Active Comparator): Non-Absorbable Sutures
  Interventions: Device: Non-Absorbable Sutures

INTERVENTIONS:
Device: Non-Absorbable Sutures — Non-Absorbable Sutures
  Arms: Non-Absorbable Suture
Device: Absorbable Suture — Absorbable suture
  Arms: Absorbable Suture

SUMMARY:
The study is to prospectively compare absorbable sutures with non-absorbable sutures used for capsular repair during hip arthroscopic procedures. Major outcomes will be measured using three questionnaires ((1) International Hip Outcome Tool-12 (iHOT-12), (2) modified Harris hip score, (3) hip outcome score) in addition to the standard of care set of 9 questionnaires. The other major outcome will be any radiographic heterotrophic ossification at the 6-month follow-up time point.

DETAILED DESCRIPTION:
1. International Hip Outcome Tool-12 is a 33-item patient-reported measure of health-related quality of life. It was designed to measure the impact of hip disease in young, active patients and to measure the effect of treatment of this disease.
2. Modified Harris hip score is composed of 8 survey questions to determine gait, functionality and pain.
3. The hip outcome score is 26 survey questions designed to asses the outcome of arthroscopic hip surgery for individuals with acetabular labral tears, including sports related questions and activities of daily living.

Standard of care questionnaires will be given at follow up clinic visits. They are the:

1. Patient Reported Outcomes Measurement Information System (PROMIS) Physical Function
2. PROMIS pain interference
3. PROMIS Global Health
4. Pain Visual Analog Scale
5. Hip Single Assessment Numeric Evaluation (SANE)
6. Modified Harris Hip Score
7. Marx Activity Scale
8. Tegner Activity Scale
9. Surgical Satisfaction

These questionnaires will be given at preoperative, 6-week, 3-month, 6-month, 1 year, 2 years and any other follow-up visits in association with surgery.

Any Radiographic images taken as standard of care (SOC) (post-operative radiographs are SOC) will be used in the study to determine Radiographic Heterotroph Ossification (HO) at 6 Months.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 18 years of age and older.
* Subject requiring surgical hip arthroscopic intervention for their hip pathology

Exclusion Criteria:

* Subjects less than 18 years of age.
* Subjects with any other medical problem precluding anesthesia or surgery.
* Unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-03-22 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
International Hip Outcome Tool-12 (IHOT-12) | Preoperative to 12 months postoperative
  12-item patient-reported measure of health-related quality of life. It was designed to measure the impact of hip disease in young, active patients and to measure the effect of treatment of this disease. Each of the 12 questions assess hip function and are scored from 0-100. 0 is a low score and 100 is high score indicating excellent function. The IHOT-12 is scored from taking the average of the 12 items of the tool and is scored 0-100, 0 being a low score and poor function and 100 being a high score indicating excellent function.
Modified Harris Hip score | Preoperative to 12 months postoperative
  composed of 8 survey questions to determine gait, functionality and pain. Each question is scored with a separate scoring range. Higher scores indicate better function and less pain. The score is calculated by adding up the assigned points for each item, dividing by the max score (91), and multiplying by 100 to create a percentage. A higher score indicates a higher level of physical function, with 100% indicating full function.
Hip Outcome Score (HOS) | Preoperative to 12 months postoperative
  28-item assessment that is divided into 2 subscales: activities of daily living (HOS-ADL;19 items) and sports-related activities (HOS-Sports;9 items).
  Of the 2 subscales, each question contains five answer choices ranging from low function (score of 0) to high function (score of 4). The maximum score possible for the HOS-ADL is 68. A high score indicates high function, and a low score indicates low function.
  The maximum score possible for the HOS-Sports is 36. A high score indicates high function, and a low score indicates low function.
  Scores for each subscale range from 0% (least function) to 100% (most function). Results can be interpreted with the following: <70 = poor result; 70-80 = fair, 80-90 = good, and 90-100 = excellent.

SECONDARY OUTCOMES:
Rate of Radiographic Heterotrophic Ossification | Evaluated at 6-months postoperatively
  Any radiographic heterotrophic ossification at the 6-month follow-up time point.

CONTACTS AND LOCATIONS:
Locations (1):
- Missouri Orthopaedic Institute, Columbia, Missouri, United States